CLINICAL TRIAL: NCT00917280
Title: Connecting the Lab to Everyday Life: The Relevance of Executive Dysfunction to Participation and Quality of Life in PD Without Dementia
Brief Title: Connecting the Lab to Everyday Life: The Relevance of Executive Dysfunction to Participation and Quality of Life in Parkinson's Disease (PD) Without Dementia
Acronym: Lab2Life
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Erin Foster, Assistant Professor of Occupational Therapy, Neurology and Psychiatry, Washington University School of Medicine
Other Study IDs: #E07-117
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease: Parkinson Disease participants without dementia
- Control: Non-PD participants, matched for age, education and gender.

SUMMARY:
The overall purpose of this research is to learn how Parkinson's disease affects thinking and memory in everyday life. Participation will involve thinking tests, questionnaires and interviews about thinking and activities in everyday life.

DETAILED DESCRIPTION:
The overall purpose of this research is to learn how Parkinson's disease affects thinking and memory in everyday life. Participation will involve thinking tests, questionnaires and interviews about thinking and activities in everyday life.

ELIGIBILITY:
Inclusion Criteria PD participants:

* WUSM Movement Disorders Clinic patients
* males or females between 40 and 70
* meet criteria for idiopathic typical PD
* classified at Hoehn & Yahr12 stage I, II, or III
* are currently treated with levodopa/carbidopa

Inclusion Criteria Control:

* The groups will be matched for age, education and gender
* No Parkinson Disease

Exclusion Criteria PD participants and Control:

* suspected dementia
* treatment with certain dopaminergic, anticholinergic or benzodiazepine medications
* other neurological problems
* brain surgery
* history or current psychotic disorder
* any condition which would interfere with testing
* control only: a biological family history of PD and being a caregiver or spouse of someone who has PD

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls:
  Recruited from community, VFH.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2008-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Foster, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States